CLINICAL TRIAL: NCT06780098
Title: KEYMAKER-U01 Substudy 01I: A Phase 2, Randomized, Umbrella Study With Rolling Arms of Investigational Agents in Participants With Previously Treated Stage IV Squamous Non-small Cell Lung Cancer (NSCLC)
Brief Title: Substudy 01I: A Study of Investigational Agents in Participants With Previously Treated Stage IV Squamous Non-small Cell Lung Cancer (NSCLC) (MK-3475-01I/KEYMAKER-U01I)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3475-01I; MK-3475-01I (Other: MSD); U1111-1314-2392 (Registry Identifier: UTN); 2024-518839-11-00 (Registry Identifier: EU CT); KEYMAKER-01I (Other: MSD)
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Lung Neoplasm
MeSH Terms: conditions — Lung Neoplasms | interventions — Docetaxel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1: Raludotatug deruxtecan (R-DXD) (Experimental): Participants receive 5.6 mg/kg of R-DXD, every 3 weeks (Q3W) (Day 1 of every 21-day cycle) via intravenous (IV) infusion until progressive disease (PD) or discontinuation.
  Interventions: Biological: R-DXD
- Arm 2: Infinatamab deruxtecan (I-DXD) High Dose (Experimental): Participants receive 12 mg/kg of I-DXD, Q3W (Day 1 of every 21-day cycle) via IV infusion until PD or discontinuation.
  Interventions: Biological: I-DXD
- Arm 3: I-DXD Low Dose (Experimental): Participants receive 8 mg/kg of I-DXD, Q3W (Day 1 of every 21-day cycle) via IV infusion until PD or discontinuation.
  Interventions: Biological: I-DXD
- Arm 4: Docetaxel (Active Comparator): Participants receive 75 mg/m^2 of Docetaxel, Q3W (Day 1 of every 21-day cycle) via IV infusion until PD or discontinuation.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Biological: R-DXD — IV Infusion
  Other Names: Raludotatug deruxtecan; MK-5909; DS-6000a
  Arms: Arm 1: Raludotatug deruxtecan (R-DXD)
Biological: I-DXD — IV Infusion
  Other Names: Ifinatamab deruxtecan; MK-2400; DS-7300a
  Arms: Arm 2: Infinatamab deruxtecan (I-DXD) High Dose; Arm 3: I-DXD Low Dose
Drug: Docetaxel — IV Infusion
  Other Names: Taxotere®
  Arms: Arm 4: Docetaxel

SUMMARY:
Researchers are looking for other ways to treat metastatic squamous non-small cell lung cancer (NSCLC). Squamous NSCLC is cancer that starts in squamous cells, which are flat cells that line the inside of the airways in the lungs. Metastatic means the cancer has spread to other parts of the body.

Standard treatment (usual treatment) for metastatic squamous NSCLC is immunotherapy with or without chemotherapy. Immunotherapy is a treatment that helps the immune system fight cancer. Chemotherapy is medicine that destroys cancer cells or stops them from growing. However, standard treatment may not work or may stop working to treat metastatic squamous NSCLC.

Researchers want to learn if study treatments that are antibody drug conjugates (ADCs) can treat metastatic squamous NSCLC that did not respond (get smaller or go away) to standard treatment. An ADC attaches to a protein on cancer cells and delivers treatment to destroy those cells.

The main goals of this study are to learn about:

* The cancer response to the study treatments compared to chemotherapy
* The safety of the study treatments and if people tolerate them

This study is one of the substudies being conducted under one pembrolizumab umbrella master protocol (MK-3475-U01/KEYMAKER-U01).

DETAILED DESCRIPTION:
The master screening protocol is MK-3475-U01 (KEYMAKER-U01) - NCT04165798

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Histologically or cytologically confirmed diagnosis of Stage IV squamous non-small cell lung cancer (NSCLC)
* Has documented disease progression per Response Evaluation Criteria In Solid Tumors 1.1 (RECIST 1.1), as assessed by investigator after receiving an anti-programmed cell death protein 1 (anti-PD-1)/programmed cell death ligand 1 (PD-L1) treatment and platinum-based chemotherapy for Stage IV disease
* Human immunodeficiency virus (HIV)-infected participants must have well controlled HIV on antiretroviral therapy (ART)
* Participants who are Hepatitis B surface antigen (HBsAg) positive are eligible if they have received Hepatitis B virus (HBV) antiviral therapy for at least 4 weeks, and have undetectable HBV viral load
* Participants with history of Hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Diagnosis of small cell lung cancer or, for mixed tumors, presence of small cell elements
* Has uncontrolled or significant cardiovascular disorder
* Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses including, but not limited to, any underlying pulmonary disorder (ie, pulmonary emboli within 3 months, severe asthma, severe chronic obstructive pulmonary disease, restrictive lung disease, pleural effusion, etc), or any autoimmune, connective tissue, or inflammatory disorders with pulmonary involvement (ie, rheumatoid arthritis, Sjogren's syndrome, sarcoidosis, etc), or prior pneumonectomy
* Participants who have adverse events (AEs) (other than alopecia) due to previous anticancer therapies must have recovered to ≤Grade 1 or baseline
* Evidence of ongoing uncontrolled systemic bacterial, fungal, or viral infection (including HIV infection)
* Has clinically significant corneal disease
* Known additional malignancy that is progressing or has required active treatment within the past 3 years
* Has known untreated central nervous system (CNS) metastases and/or carcinomatous meningitis
* Evidence of any leptomeningeal disease
* History of (noninfectious) pneumonitis/Interstitial Lung Disease (ILD) that required steroids or has current pneumonitis/ILD, and/or suspected ILD/pneumonitis
* Active autoimmune disease that has required systemic treatment in the past 2 years. Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid) is allowed
* Active infection requiring systemic therapy
* HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease
* Active inflammatory bowel disease requiring immunosuppressive medication or previous clear history of inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis, or chronic diarrhea)
* Known history of, or active, neurologic paraneoplastic syndrome
* History of allogeneic tissue/solid organ transplant
* Has not adequately recovered from major surgery or have ongoing surgical complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2032-03-02 (Estimated); Study Completion 2032-03-02 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 81 months
  ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) as assessed per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1). ORR will be assessed by Blinded Independent Central Review (BICR). The percentage of participants who experience CR or PR as assessed by the investigator will be presented.
Number of participants who experience one or more adverse events (AEs) | Up to approximately 81 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be reported.
Number of participants who discontinue study intervention due to an AE | Up to approximately 81 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study treatment due to an AE will be reported.

SECONDARY OUTCOMES:
Duration of Response (DOR) | Up to approximately 81 months
  For participants who demonstrate a confirmed CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until PD or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR as assessed by BICR will be presented.
Progression-free Survival (PFS) | Up to approximately 81 months
  PFS is defined as the time from randomization to the first documented PD or death due to any cause, whichever occurs first as assessed by (RECIST 1.1). PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by BICR will be presented.
Overall Survival (OS) | Up to approximately 81 months
  OS is defined as time from randomization to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (37):
- United States (2):
  - University of Kentucky Chandler Medical Center ( Site 0019), Lexington, Kentucky
  - MedStar Franklin Square Medical Center ( Site 0033), Baltimore, Maryland
- Chile (3):
  - Centro de Estudios Clínicos SAGA ( Site 0161), Santiago, Region M. de Santiago
  - FALP ( Site 0160), Santiago, Region M. de Santiago
  - Bradfordhill ( Site 0162), Santiago, Region M. de Santiago
- China (7):
  - Chongqing University Cancer Hospital ( Site 0304), Chongqing, Chongqing Municipality
  - Fujian Provincial Cancer Hospital ( Site 0310), Fuzhou, Fujian
  - Guangxi Medical University Cancer Hospital ( Site 0303), Nanning, Guangxi
  - Henan Cancer Hospital ( Site 0311), Zhengzhou, Henan
  - Nanjing Drum Tower Hospital JiangBei International Branch Hospital ( Site 0309), Nanjing, Jiangsu
  - Shanghai Chest Hospital ( Site 0308), Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital ( Site 0300), Shanghai, Shanghai Municipality
- Germany (2):
  - UniversitaetsklInikum Tuebingen ( Site 0192), Tübingen, Baden-Wurttemberg
  - Charite-Universitaetsmedizin Berlin ( Site 0191), Berlin
- Greece (2):
  - THORACIC GENERAL HOSPITAL OF ATHENS "I SOTIRIA" ( Site 0204), Athens, Attica
  - European Interbalkan Medical Center-Oncology Department ( Site 0205), Thessaloniki
- Hungary (3):
  - Bacs-Kiskun Varmegyei Oktatokorhaz ( Site 0063), Kecskemét, Bács-Kiskun county
  - Petz Aladar Egyetemi Oktato Korhaz ( Site 0062), Győr, Győr-Moson-Sopron
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Gyula Korhaz-Rendelointezet ( Site 0061), Szolnok, Jász-Nagykun-Szolnok
- Israel (6):
  - Rambam Health Care Campus ( Site 0076), Haifa
  - Shaare Zedek Medical Center ( Site 0075), Jerusalem
  - Meir Medical Center ( Site 0071), Kfar Saba
  - Rabin Medical Center ( Site 0074), Petah Tikva
  - Sheba Medical Center ( Site 0070), Ramat Gan
  - Sourasky Medical Center ( Site 0077), Tel Aviv
- Italy (4):
  - Azienda Ospedaliera Universitaria Careggi ( Site 0173), Florence
  - Ospedale San Raffaele. ( Site 0171), Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori ( Site 0175), Milan
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore ( Site 0174), Roma
- Poland (4):
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii ( Site 0153), Poznan, Greater Poland Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie ( Site 0151), Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne-Early Clinical Trials Unit ( Site 0150), Gdansk, Pomeranian Voivodeship
  - Szpital Wojewódzki im. Mikoaja Kopernika w Koszalinie ( Site 0152), Koszalin, West Pomeranian Voivodeship
- Spain (2):
  - Hospital Clinic de Barcelona ( Site 0092), Barcelona
  - Hospital Universitario Quiron Madrid ( Site 0091), Madrid
- Turkey (Türkiye) (2):
  - Hacettepe Universitesi Tip Fakultesi Hastanesi ( Site 0140), Ankara
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi ( Site 0144), Istanbul

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com